CLINICAL TRIAL: NCT02514317
Title: Ultrasound-assisted Percutaneous Release of Carpal Tunnel Syndrome
Brief Title: Percutaneous Treatment of Carpal Tunnel Syndrome With Scan
Acronym: ECHOCARPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-058
Record Dates: First submitted 2015-07-23; First posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- percutaneous treatment (Experimental): percutaneous treatment of carpal tunnel syndrome under ultrasound guidance in interventional radiology room.
  Interventions: Procedure: percutaneous treatment; Device: Ultrasound

INTERVENTIONS:
Procedure: percutaneous treatment
Device: Ultrasound

SUMMARY:
The objective of the study is to evaluate in patients suffering from carpal tunnel syndrome resistant to medical treatment, clinical course after percutaneous treatment under ultrasound guidance. 40 patients will be included in the study. The following parameters will be evaluated: patient satisfaction, pain, functional disability, quality of life and time to return to work. The medico-economic aspect will be analyzed.

DETAILED DESCRIPTION:
Ultrasound analysis of Carpal tunnel is used for many years, especially for diagnostic purposes. Investigators have shown, first by a study of 104 cadavers that it was possible to reduce the opening by making the gesture under ultrasound guidance and to perform the procedure under local anesthesia. Then investigators performed an open study of 25 patients confirming the absence of iatrogenic lesions with this new technique.

The percutaneous treatment of carpal tunnel syndrome under ultrasound guidance is a gesture of interventional radiology. One can envisage making this type of treatment in interventional radiology room which overcomes the operating room and thus reduce costs.

The objective of the study is to continue the study of percutaneous treatment of carpal tunnel syndrome under ultrasound guidance by an open study conducted in interventional radiology room.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years who signed the informed consent.
* Patient with an Carpal Tunnel Syndrome

Exclusion Criteria:

* patient has already undergone surgery of Carpal Tunnel Syndrome
* Patient with contra-indications to anesthesia (heart failure, kidney, liver).
* Pregnant women
* alcoholics in weaning period
* Patient whose consent is altered or unable to get a safety procedure
* Patient with contra-indication to lidocaine
* Patient with contra-indication for the realization of ultrasound endoscopy (carpal tunnel syndrome secondary or anastomosis between the median and ulnar nerves: anastomosis Berritini)

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain (visual analogic scale) | change between baseline and day 90 after surgery
  visual analogic scale
paresthesia | change between baseline and day 90 after surgery
muscle strength (dynamometer JAMARD) | change between baseline and day 90 after surgery
  dynamometer JAMARD

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Caen, France